CLINICAL TRIAL: NCT00204828
Title: T Regulatory and Childhood Asthma
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: H-2004-0224; R01HL080072 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Childhood Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, PBMC culture supes and nasal lavage
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1.: Children with asthma
- 2.: Children without asthma

SUMMARY:
This is an epidemiologic study, examining environmental exposures and affect on immune development.

DETAILED DESCRIPTION:
This is an epidemiologic study, examining environmental exposures and affect on immune development. The study has completed enrollment

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe asthma

Exclusion Criteria:

-

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 6-7 yo children of either gender
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2005-10; Primary Completion 2007-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Childhood asthma | 3 years
Allergic sensitization | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: James Gern, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No